CLINICAL TRIAL: NCT07209774
Title: Healthspan Connect Programme of Research
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer Research UK (Other); French National Cancer Institute (Institut National Du Cancer - France) (Unknown); Bowelbabe Fund (Unknown); Republique Francaise (Unknown)
Responsible Party: Sponsor
Other Study IDs: 362403; 1OT2CA297289-01 (NIH)
Record Dates: First submitted 2025-09-26; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Mental Health; Ageing Well; Resilience; Cognitive Health; Psychological Health; Environmental Health Effects; Cardiovascular Health; Metabolic Health; Neurological Health; Musculoskeletal Health; Respiratory Health; Allergies; Eye Health; Other
Keywords: Healthy ageing; Healthspan; Longevity; Ageing resilience; Life course determinants; Multiple long-term conditions; Digital health research; Remote monitoring; Mobile health (mHealth); Wearables; Biobank; Biological specimen collection; Home-based sample collection; Epidemiology; Longitudinal cohort study; Adolescents and ageing; Underrepresented populations in research; Behaviour change; Environmental exposures; Data linkage; Electronic health records (EHR); United Kingdom
MeSH Terms: conditions — Neoplasms; Psychological Well-Being; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthspan Connect is a new research programme designed to understand what helps people stay healthy as they age. The programme will explore how lifestyle, environment, genetics, and social factors influence healthy ageing and overall wellbeing.

The programme will recruit participants aged 12 years and older across the UK. By including adolescents, the programme aims to understand how early life behaviours and experiences shape long-term health. There is no upper age limit, and people from all backgrounds are encouraged to participate. Special pathways ensure that young participants provide consent in an age-appropriate way.

Healthspan Connect is a digital and home-based study, meaning participants can take part from home using smartphones, computers, and online surveys. Participants may also be asked to collect samples such as blood, saliva, stool, urine, or other biological specimens at home using easy-to-use kits. In some sub-studies, participants may be invited to attend research visits for additional tests, scans, or clinical assessments. Family members and close contacts may also be invited to participate in some studies.

Through Healthspan Connect, researchers aim to:

* Identify the biological, environmental, and social factors that help people live longer, healthier lives.
* Understand how different groups, including those historically underrepresented in research, experience ageing.
* Explore ways to support behaviour changes that improve health over the lifespan.
* Provide near real-time information to inform health policies and interventions.

Participants may also be asked for permission to link their information with health records, education records, and environmental data to better understand health outcomes over time.

This programme will serve as a flexible platform for multiple sub-studies, allowing participants to contribute to a wide range of research questions related to healthy ageing, resilience, and long-term health. All data and biological samples will be stored securely and used to advance scientific knowledge, with participant privacy carefully protected.

DETAILED DESCRIPTION:
1. **SUMMARY**

**a) Rationale**

Healthspan Connect is a new Programme of Research aimed at understanding the life course determinants of healthy lifespan and gain real--time epidemiological insights into health--policy relevant questions.

Healthspan Connect will study healthy volunteers and use digital and remote methods to support healthspan and ageing research, as well as study multiple long-term conditions. The study builds from the ZOE Health study, which Steves designed, with a view to creating capability for rapid scientific answers to policy driven research questions and will also be guided in part by CARICE (Centre for Ageing Resilience in a Changing Environment), a KCL-led research and policy centre on ageing resilience directed by Steves. Healthspan Connect, which will be a vehicle for agile research and the programme sub-studies preferentially focussed on answering clinically and policy relevant research questions.

Healthy ageing and an extended health span are essential as they directly impact quality of life, individual well-being, and societal sustainability. With populations ageing globally, the objective is not only to increase life expectancy but to ensure that these additional years are lived in good health, free from chronic diseases and disabilities. A longer health span enables individuals to maintain their independence, continue contributing to their communities, and enjoy a better quality of life in their later years. Moreover, promoting healthy ageing alleviates the strain on healthcare systems and social care, which can become overburdened by the rising incidence of age-related diseases. By prioritising healthy ageing, this research aims to enhance overall life satisfaction, reduce healthcare costs, and foster more resilient societies where older adults remain active, engaged, and healthy for as long as possible. Additionally, it is crucial to involve underrepresented populations in ageing research to ensure that the benefits of health span extension are equitably distributed. Understanding how ageing and health resilience manifest in diverse groups, including those historically under-represented in research, will enable the development of more inclusive public health strategies and interventions that address the needs of all individuals as they age.

Involving participants between the ages of 12 and 15 years will enable the study to capture early determinants of healthy ageing by following participants from adolescence to adulthood. This approach allows for the observation of physical, cognitive, and mental health trajectories from a critical developmental stage, when many lifelong health behaviours are established and when the risk of onset for certain health conditions begins to emerge. Adolescents remain underrepresented in longitudinal studies, yet their inclusion is essential for understanding how early life experiences, social environments, and behavioural patterns contribute to ageing outcomes. Following individuals from their teenage years will enhance the cohort's representativeness, support trans-generational analyses, and provide unique insights into how contemporary influences shape lifelong health and wellbeing.

Healthspan Connect is a new longitudinal cohort dedicated to researching ageing and health resilience. Healthspan Connect will enable advancements in study design, methodology and large--scale data collection through remote participant recruitment, mobile health data capture via connected devices and apps, and the ability to collect samples remotely. The research programme will focus on strategies to maximise the number of years individuals spend in good health by exploring the underlying mechanisms of health resilience. This will involve investigating the biological, environmental and social factors that contribute to ageing and how these can be influenced to promote health. Additionally, the programme will place a strong emphasis on including underrepresented groups to ensure that the findings are inclusive and applicable to diverse populations. The research will also address prevention and early detection, with the cohort serving as a dynamic resource for studying these factors over time. Furthermore, the programme will provide participants with insights into their health and the potential impact of various risk factors. Alongside this, the research will delve into the drivers and barriers of behaviour change, aiming to understand how individuals can be supported in making lifestyle changes that enhance their health span. This comprehensive approach will provide valuable insights that will inform strategies and public policies to support longevity, health resilience, and effective behaviour change across all segments of society.

**b) Expanding Research Access**

Digital platforms have become integral to modern health research and clinical trials, offering a range of functionalities that enhance the agility and ability of research teams to conduct studies more efficiently. For instance, the ZOE COVID Symptom Study recruited over four million users through a mobile app, enabling ZOE and researchers at KCL to monitor the spread of COVID-19, identify risk factors, and predict outbreaks based on self-reported symptoms. Similarly, the COVID-19 Citizen Science Study used the Eureka Research Platform to recruit over 50,000 participants, collecting real-time, self-reported health data via digital surveys, with a sustained engagement rate of around 59% every four weeks. The unprecedented scale and speed of data collection during a pandemic demonstrates how digital platforms can extend the reach of research beyond traditional settings. Tools such as remote recruitment, e-consent, app-based data collection, geofencing, and digital interventions allow researchers to respond rapidly to emerging challenges while increasing inclusivity.

One of the most significant advantages of digital platforms is their ability to engage under-researched and underserved populations. By removing geographical and logistical barriers, these platforms can involve individuals who might otherwise be excluded due to health limitations, social barriers, or lack of access to major research centres. For example, studies have shown that digital tools can improve representation by enabling participation from people across different socioeconomic backgrounds, age groups, and ethnic communities. Furthermore, the use of intelligent systems for participant matching and onboarding increases the ability to tailor recruitment efforts towards populations that have historically been underrepresented in clinical research. The collection of real-world data through wearables and mobile apps also supports a more patient-centred approach, capturing insights from everyday life that are often missed in clinic-based studies. Despite challenges such as digital literacy and internet access, digital platforms are helping to reshape clinical research into a more agile, inclusive, and representative endeavour.

To expand research access and ensure that younger people can contribute meaningfully, the study is designed to include participants from the age of 12, with two tailored consent pathways for 12 to15-year-olds. The adult-initiated pathway enables a parent or guardian who is already a volunteer to invite their child to take part, while the child-initiated pathway allows a young person to express interest themselves, with parental consent then sought. In both pathways, comprehension checks are built in to confirm the young person understands the study before consent is finalised. This approach is consistent with the UN Convention on the Rights of the Child (UNCRC), balancing autonomy and protection, and removing unnecessary barriers to participation for this underrepresented age group.

**c) Participant Support**

Of the current application, the participant advisory group for the COVID Symptom Study (CSS) Biobank (20/YH/0298) were consulted in July 2025 about the Healthspan Connect Programme of Research model and all members present were supportive of the new model and agreeable to be invited to sub-studies in this way. Additionally, a survey conducted in April 2024 among participants in the CSS Biobank asked whether they would be interested in taking part in similar studies beyond COVID-related research. Of the respondents, 3,242 (97%) indicated that they 'may' or 'definitely would'. This highlights the strength of the digital platform and study design in keeping participants engaged, making it a valuable foundation for future research efforts.

This current REC application describes Healthspan Connect as a Programme of Research, alongside an application for a Research Tissue Bank (Healthspan Connect Biobank) which will act as a biorepository for the Programme of Research, allowing it to also be a valuable resource for the wider scientific community.

**d) Aims and objectives**

Healthspan Connect aims to:

1. Investigate the biological, environmental, and social factors that contribute to healthy ageing and health resilience. This will involve a comprehensive analysis of how these factors interact and can be influenced to maximise the number of years individuals spend in good health.
2. Ensure the inclusivity and representativeness of the research by actively involving underrepresented populations. The aim is to generate findings that are applicable across diverse groups, enabling the development of public health strategies and interventions that are equitable and effective for all segments of society.
3. Provide participants with insights into their health and study the drivers and barriers to behaviour change. This will include offering insights into health risks and understanding how to effectively support individuals in adopting behaviours that enhance their health span, ultimately informing strategies and public policies that promote longevity and health resilience.
4. Be an agile platform to answer policy relevant questions as and when they arise to provide near real-time data for policymakers and the public. Envisaged uses include analysis of effects of local and national health policy interventions (e.g. changes in fortification of food, emissions zoning, neighbourhood health services) and environmental changes (climate change, seasonal variations, new infectious diseases).

**e) Proposed cohort**

Healthspan Connect will recruit participants that have taken part in previous studies health studies linked to The Department of Twin Research and collaborating organisations. They will subsequently be able to join sub-studies under this Programme of Research model. Any biological samples collected as part of Healthspan Connect will be stored in the Healthspan Connect Biobank, linked to this application.

2. **METHODS**

**a) Programme design**

The Healthspan Connect Programme of Research will enable us to collect data and samples longitudinally from participants who take part in specific sub-studies, funded by grant programmes or by access requests from external collaborators. According to sub-study specific designs, researchers will collect biological specimens and/or data from Healthspan Connect participants mainly through home-based or postal studies. Researchers may ask participants to attend research visits for certain sub-studies. Researchers will recall participants at follow up time points to update their baseline data and to donate additional specimens as required by sub-study protocols.

**b) Recruitment to the programme**

Participants will be eligible to join Healthspan Connect if they are currently resident in the UK and are 12 years or older. Participants will be made aware of Healthspan Connect through media coverage, flyers and posters in public settings, social media campaigns, recruitment campaigns, partnerships with the NHS, community groups and health companies such as ZOE, and word of mouth from existing volunteers.

**c) Eligibility to join Healthspan Connect**

To join Healthspan Connect, prospective participants must be at least 12 years old, resident in the United Kingdom, and able to participate in Healthspan Connect online (computer or smartphone). There is no upper age limit. Participants must be able to provide informed consent and complete digital questionnaires independently. Participants aged 12-15 years old must provide parent/guardian consent to take part.

**d) Recruitment to substudies within the programme**

Once included in the Healthspan Connect programme, participants will be able to take part in sub-studies run by collaborators within the programme. This may include collecting biological specimens and health or lifestyle-related information at home or at their local medical centre and returning the specimens by post or completing questionnaires. Participants may also be invited to come in for research visits at the DTR or partner organisations.

The programme will recruit participants to Healthspan Connect via an online platform. Potentially eligible participants will be invited to self-enrol in sub-studies in line with the eligibility criteria and recruitment protocol for each sub-study. Participants will be able to take part in multiple sub-studies, subject to eligibility.

The programme may invite participants' family members and household members to take part in sub-studies. The programme may also invite close contacts of participants to enable recruitment of hard to reach populations. This will be done through contact with the participant first, to ensure researchers may reach out to the close contact/family/household members. The programme will recruit family/household members or close contacts by telephone, email or letter to donate selected biological specimens and may ask them to complete questionnaires. Biological specimens and health or lifestyle related information will be collected at home, at the family/household member's or close contacts local medical centre, or partner organisation and returned by post. The programme may also invite family/household members or close contacts to attend visits depending on the nature of the tests they are asked to take part in.

Each sub-study will have its own Participant Information Sheet (PIS).

Participants will be made aware of what will happen when recruited to a specific substudy, the tests that will take place, the specimens that will be collected, any risks associated, and any results that may be provided. The prospective participants will also have an opportunity to ask questions via online platforms, email or over the phone and discuss any issues they may be concerned with.

**e) Biological specimen and data collection**

Participants may be invited to contribute the following specimens and data through the programme and future sub-studies:

* Questionnaires
* Paper-based, or collected through secure platforms such as Qualtrics or REDCap
* Self-collected biological samples such as capillary blood, urine, stool, saliva, sweat, nail, hair and semen
* Collected by participants themselves with little or no supervision required, through easy-to-use kits and instructions
* Environmental samples such as local drinking water, soil or dust, or local environmental sensors, such as air quality/temperature/noise
* Cognitive and psychological tests
* Delivered through online programmes such as Cognitron, CANTAB, or in person by trained staff e.g. verbal fluency
* Using apps, wearables, or smart clinical devices (e.g. continuous glucose monitors or fitness trackers) to record, monitor and track measures such as diet, health, sleep, mood, exercise and environmental information such as location or pollution
* Focus groups and interviews
* Either in person, online or over the phone
* Clinical scans and imaging such as MRI, ultrasound, DXA and EEGs
* Performed by trained staff and with clinician support where required
* All local safety protocols in effect
* Other imaging such as photographs and fingerprints
* Other types of digital footprints such as loyalty cards
* Clinical assessments and tests such as height, weight, blood pressure, fitness tests, skin assessments, dental and oral assessments, allergy testing, eye tests, hearing tests, taste tests and other sensory tests e.g. temperature
* Biological samples collected by trained staff, such as venous blood and tissue samples through biopsies e.g. fat, muscle
* Venous blood collection and cannulation performed by staff trained in phlebotomy
* Biopsies performed by staff trained in the relevant biopsy method
* Lifestyle and/or dietary changes, including
* dietary supplements
* pre/probiotics
* following a prescribed or standardised diet
* meal challenges
* other interventions that do not involve the use of medical treatments, for example, eye drops or local anaesthetic

Biological specimens will primarily be collected through postal studies, whereby participants will be provided with easy-to-use kits and instructions. We will provide details about any home collection or postal specimens in specific VIS for each sub-study. The programme may also arrange for visits to take place at partner organisations or collaborating centres or invite participants to have samples collected through a partner organisation. The programme may also from time to time undertake home visits to allow participants to continue to take part in Healthspan Connect research if they are unable to attend in person.

Biological specimens and data from family members will primarily be collected by post unless specific sub-studies require participants to attend a research visit. Researchers will issue packs for any specimens that need to be collected before the visit and brought to the collaborating centres, such as faecal specimens, urine or saliva.

Data collected from participants and derived from their biological specimens will include phenotypic data from self-reported questionnaires or from collaborative sources, sequenced data (Genotyping, Whole Genome Sequencing), omics data and analysed or derived datasets from internal and collaborative analysis.

Questionnaire data will be collected using online questionnaires. Questionnaires will be provided in English, but in the future may be offered in other languages and translated to facilitate participation from hard-to-reach groups.

**f) Records linkage**

Upon signing up to Healthspan Connect, researchers will ask participants permission to request additional information about them through linkage to past, current and future records held by the NHS, government bodies or other trusted organisations. For example, researchers will ask permission to link to participants' electronic healthcare records available through the NHS and their GP; education records held by the Department for Education; and environmental records such as information held by organisations such as the ONS or Centre for Hydrology and Ecology based on postcodes. Once appropriate data sharing agreements are in place, researchers request data by securely providing identifiers to the data holders. Data received back is then integrated with our existing data within a secure environment. The programme may also link to participants' data through other data sharing and linkage infrastructure, for example the UK Longitudinal Linkage Collaboration (UK LLC). The programme may also invite participants to allow it to link to their retail loyalty card data (e.g. Nectar cards or Boots Advantage cards).

*Health record linkage and the UK LLC*

Health record data linkage is performed to enhance the depth, breadth, and usefulness of Healthspan Connect study data by combining study data with information from health records to generate a more comprehensive understanding of health outcomes over time.

Healthspan Connect will apply to join the UK Longitudinal Linkage Collaboration (UK LLC) to facilitate the health record data linkage process. Within the UK LLC, trusted third parties are responsible for linking data from sources such as DCHW and NHS England to ~~CSS Biobank~~ data. Once linked, the data would be made available to approved Healthspan Connect researchers through a secure access process.

As part of the arrangement with the UK LLC, Healthspan Connect would become one of the UK LLC's Longitudinal Population Studies (LPS). Healthspan Connect data necessary to conduct health data linkage would be integrated into the UK LLC's Trusted Research Environment (TRE). Researchers interested in accessing Healthspan Connect data from the UK LLC would need to apply directly through the Healthspan Connect study's own data access procedures (see section 3k) to ensure appropriate use in accordance with the study data sharing policy and participant consent.

**g) Data analysis**

Initial reception and processing of biological specimens will take place at the DTR laboratory facility at the Rayne Institute, KCL, St Thomas' Hospital campus. Some specimens are sent to pathology labs at Guys & St Thomas' Hospital. All other specimens will be processed for long-term storage (see Section 3h). Analysis of biological specimens to generate data for research projects will be undertaken by each specific research team, either internally at the DTR or externally at other institutions under appropriate data transfer agreements.

Quality control (QC) and quality assurance (QA) processes will be followed to ensure data integrity. Metadata will then be assigned to all questionnaire data.

3. **PROSPECT UK (first Healthspan Connect sub-study)**

PROSPECT-UK is a UK-based prospective longitudinal cohort study designed to investigate dietary, lifestyle, and other health-related risk factors associated with early-onset colorectal cancer (EOCRC), defined as colorectal cancer diagnosed before age 50. Participants will initially be recruited from existing longitudinal cohorts, with baseline data collected on diet, lifestyle behaviours, medical history, and anthropometric measures. Annual follow-up questionnaires will capture changes in exposures over time. Electronic health record (EHR) linkage will be used to identify incident cases of EOCRC and colorectal adenomas. A subsample of participants may provide biological specimens, including blood and stool, to enable nested case-control studies and mechanistic analyses.

The primary objective is to identify and quantify associations between diet, lifestyle, and health-related risk factors and the development of EOCRC and its precursors. Secondary objectives include establishing a longitudinal cohort for ongoing EOCRC research, facilitating future nested studies, and supporting mechanistic investigations using collected biospecimens.

The study will generate high-quality, longitudinal data on EOCRC risk factors in a UK population, addressing current gaps in knowledge and supporting evidence-based prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years or older at time of enrollment.
* Resident in the United Kingdom.
* Able to participate in the study using digital tools (smartphone, tablet, or computer).
* Able to provide informed consent (digital consent accepted).
* For participants aged 12-15 years: must have parent/guardian consent in addition to their own assent.

Exclusion Criteria:

* Individuals unable to provide informed consent (or parental consent where applicable).
* Individuals not resident in the UK.
* Individuals unable to complete study requirements due to lack of internet access, inability to use digital devices, or severe digital literacy barriers.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit a large, diverse population of UK residents aged 12 years and older, including adolescents, young adults, and adults across the life course. Participants will be drawn from the general population through open digital recruitment methods and will not be limited by specific disease status. The cohort aims to reflect the socioeconomic, geographic, and ethnic diversity of the UK, with particular efforts to include groups typically underrepresented in health research.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2056-01-05 (Estimated); Study Completion 2056-01-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of early-onset colorectal cancer (EOCRC) | Through study completion, anticipated ≥10 years
  Primary outcome for the first sub-study under the Healthspan Connect programme of research (PROSPECT UK). Defined as a new diagnosis of colorectal cancer before age 50. Confirmed via data from Electronic Health Record Linkage.
Incidence of early-onset colorectal adenoma (EOCA) | Through study completion, anticipated ≥10 years
  Primary outcome for the first sub-study under the Healthspan Connect programme of research (PROSPECT UK). Defined as a new diagnosis of colorectal adenoma before age 50. Confirmed via data from Electronic Health Record Linkage.